CLINICAL TRIAL: NCT02643160
Title: Analyzing the Effect of Functional Trunk Training on Upper and Lower Limb Motor Function in Children With Spastic Cerebral Palsy
Brief Title: Analyzing the Effect of Trunk Training on Limbs in Children With Spastic Cerebral Palsy
Acronym: FTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GO 14 135
Record Dates: First submitted 2015-11-25; First posted 2015-12-31 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Cerebral Palsy, Spastic
Keywords: Trunk Training; Motor Function
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Functional Trunk Training Group (Experimental): Functional Trunk Training which includes strengthening of trunk muscle and functional activities including trunk region.
  Interventions: Other: Functional Trunk Training
- Control Group (No Intervention): No intervention, the continued their regular physical therapy

INTERVENTIONS:
Other: Functional Trunk Training — The intervention includes neurodevelopment treatment, muscle strengthening and functional activities of trunk region
  Arms: Functional Trunk Training Group

SUMMARY:
The purpose of this study is to analyze if trunk training has effects on trunk, upper, lower extremity motor functions in children with spastic Cerebral Palsy. Second purpose is to analyze the relation between trunk control and prematurity, birth weight, upper and lower extremity motor functions in children with spastic Cerebral Palsy.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is a condition caused by a lesion occurred in immature brain during prenatal, natal or postnatal period. Children with CP may have motor, cognitive, sensory, auditory, behavioral problems during their lifespan. Spastic type CP is most common type of CP and many children with spastic CP have both trunk and limb impairment. Physiotherapy is very important for improving motor function and protect from secondary impairments in this children and should start as early as possible. The aim of this study is to analyze if trunk training has effects on trunk, upper and lower extremity motor function in children with spastic CP. 38 children with spastic CP between 4-18 years age are included in this study. Both genders are included. The Participants randomized according to their gross motor function classification system levels and their age. Before intervention all groups assessed with assessment tools which assess muscle spasticity, balance, gross motor function, trunk control and walking characteristics. After randomization there wasn't any intervention for control group; they continued their regular physiotherapy in special education centers two times a week. Study group received trunk training two times a week in addition to their regular physiotherapy in special education centers during 8 weeks. After 8 weeks all groups assessed with the same assessment tools.

ELIGIBILITY:
Inclusion Criteria:

1. Children with spastic cerebral palsy effected bilaterally
2. Between 4-18 years age

Exclusion Criteria:

1. Received orthopedic surgery during last 6 weeks
2. Receive Botulinum Toxin injection during last 6 weeks
3. Mentally retarded children with communication limitations
4. Had epileptic seizures during last 12 moths -

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2014-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in trunk control over time assessed with Trunk Control Measurement Scale. | At baseline and 8 weeks after baseline
  Assessing change in trunk control

SECONDARY OUTCOMES:
Change in daily living activities and participation over time assessed with Child Health Questionary Parent Form 50. | At baseline and 8 weeks after baseline
  Assessment of child's daily living activities and participation
Change in muscle activation over time assessed with Surface Electromyography. | At baseline and 8 weeks after baseline
  Assessment of muscle activation
Change in muscle spasticity over time assessed with Modified Tardieu Scale. | At baseline and 8 weeks after baseline
  Assessing muscle spasticity
Change in gross motor function over time assessed with Gross Motor Function Measurement | At baseline and 8 weeks after baseline
  Assessing gross motor function
Change in upper extremity skills over time assessed with Quality of Upper Extremity Skills Test | At baseline and 8 weeks after baseline
  Assessing upper extremity skills
Change in loco motion over time assessed with Gillette Functional Assessment Scale | At baseline and 8 weeks after baseline
  Assessing loco motion.
Change in walking parameters over time assessed with Physicians Rating Scale | At baseline and 8 weeks after baseline
  Assessing walking parameters
Change in functional loco motion over time assessed with Timed Up and Go Test | At baseline and 8 weeks after baseline
  Assessing functional loco motion
Change in walking speed over time assessed with 1 Minute Walk Test | At baseline and 8 weeks after baseline
  Assessing walking speed
Change in balance over time assessed with Pediatric Balance Scale | At baseline and 8 weeks after baseline
  Assessing balance
Change in impact of having a disabled child on family over time assessed with Impact on Family Scale | At baseline and 8 weeks after baseline
  Assessing impact on family to have a disabled child
Change in independence level over time assessed with Functional Independence Measure for Kids | At baseline and 8 weeks after baseline
  Assessing independence level

CONTACTS AND LOCATIONS:
Overall Officials: Mintaze KEREM GÜNEL, Professor, Study Director — Hacettepe University, Graduate School of Health Sciences, Physical Therapy and Rehabilitation Department

REFERENCES:
- [Result] Heyrman L, Molenaers G, Desloovere K, Verheyden G, De Cat J, Monbaliu E, Feys H. A clinical tool to measure trunk control in children with cerebral palsy: the Trunk Control Measurement Scale. Res Dev Disabil. 2011 Nov-Dec;32(6):2624-35. doi: 10.1016/j.ridd.2011.06.012. Epub 2011 Jul 14. PMID 21757321